CLINICAL TRIAL: NCT05128370
Title: Visual Observation Scale for the Upper Limb During Walking in Patients After Stroke.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Algemeen Ziekenhuis Maria Middelares (Other); Belgisch Zee Instituut Oostende (Unknown)
Responsible Party: Sponsor
Other Study IDs: BC-10309
Record Dates: First submitted 2021-10-25; First posted 2021-11-22 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2021-10

CONDITIONS: Gait, Hemiplegic; Stroke; Upper Extremity Paresis
Keywords: arm swing; visual observation
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke; Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke group: Stroke patients who can walk independently for at least 10 meters without rest. Unilateral walking aids are allowed.
  Interventions: Other: Visual observation of arm swing during walking

INTERVENTIONS:
Other: Visual observation of arm swing during walking — The gait pattern of the stroke patients will be scored based on a visual observation scale. Additional components concerning the arm swing have been added to an existing scale.

SUMMARY:
For several years now, it has been demonstrated that the upper limb plays an important role in the function of an efficient and balanced gait pattern in healthy adults. After a stroke, the reduced muscle strength has a clear influence on the gait pattern, but also on the active movement possibilities of the upper limb. However, the role of the upper limb during gait is not sufficiently explored in the literature. The gold standard for motion analysis is a 3D analysis performed with infrared cameras capturing reflective markers during gait. Unfortunately, it is not possible for all people after a stroke to undergo this examination. On the one hand, patients must already have a certain degree of independence with regard to gait. On the other hand, not all centers have access to this expensive accommodation. There are some validated observation scales for people after stroke to describe the gait based on a 2D video image. This method is much more accessible and can be applied by any therapist. However, to date there has been little attention paid to the upper limb in these observation scales. Therefore, analogous to the observation scales for gait, an observation scale for the upper limb during gait was set up. The use of this scale can add value to the rehabilitation of people after a stroke.

* The treatment team will receive information about the patient's complete movement pattern.
* The arm will be more prominent when setting rehabilitation goals related to gait. This can lead to a positive effect on the gait pattern itself, but also to more attention being paid to the arm, which has a more difficult recovery than the leg after a stroke.

The aim of the current study will be

* to determine the inter and intra tester reliability of this visual observation scale
* to investigate if the results of the visual observation scale correlate to a 3D assessment performed in a subgroup of participants

DETAILED DESCRIPTION:
Patients will be walking for 4x10 m. During this walking a 2D video recording in the frontal (back and front view) and sagittal plane (left and right sided view) will be performed.

Supervision of therapist during walking is allowed. Therapist cannot help the patient during walking.

This images will be used to score the visual observation scale (G.A.I.T) and the additional observation scale developed for this study.

In a subgroup of participants from the Ghent University Hospital, a 3D assessment will be made on an instrumented treadmill (GRAIL, Motek), which will be used as a golden standard to compare with.

Additional clinical parameters will be investigated to describe the study group.

ELIGIBILITY:
Inclusion Criteria:

* All stroke patients who are able to walk with or without the use of a unilateral walking device (stick, tripod) for at least 10 m.
* Normal ambulation prior to stroke.
* Unilateral stroke.

Exclusion Criteria:

* Other neurologic conditions.
* Orthopedic conditions that influence gait.
* Visual impairments that impede independent walking.
* Cerebellar stroke

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patient from inpatient or outpatient rehabilitation centers.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Interrater reliability of the upper limb observation scale | Single point of assessment within one week after the 2D video has been made
  Intraclass correlation coefficient between the different raters who rate the same observation at the same time.
Intrarater reliability of the upper limb observation scale | Assessment at 2 points in time with an interval of 2 weeks.
  Intraclass correlation coefficient between the same rater rating the videos within a period of 2 weeks from each other.
Kinematic assessment of the arm swing during walking | Single point of assessment within one week
  Correlation statistics between items of the upper limb observation scale and kinematic graphs of the 3D assessment which will be performed within a week after the 2D assessment.
Visual observation scale for the upper limb during walking | Single point of assessment within one week after the 2D video has been made
  Total score on the upper limb visual observation scale (max score 34)

SECONDARY OUTCOMES:
Demographic variables | Single point of assessment at assessment day 1
  Age, gender, date of birth, stroke date, type of stroke, side of paresis, stroke location
Fugl Meyer assessment upper limb section | Single point of assessment at assessment day 1
  Active recovery of the upper limb
Fugl Meyer assessment lower limb section | Single point of assessment at assessment day 1
  Active recovery of the lower limb
Upper limb spasticity (Modified Ashworth Scale) | Single point of assessment at assessment day 1
  Modified Ashworth Scale (minimum 0 - maximum 4, higher score is more spasticity = worse outcome) of shoulder flexors, extensors, internal rotators, external rotators, adductors, abductors, elbow flexors, elbow extensors, wrist flexors, wrist extensors, finger flexors and finger extensors
Passive range of motion shoulder and elbow | Single point of assessment at assessment day 1
  Goniometric measurement of shoulder flexion, abduction, external rotation, internal rotation and elbow flexion/extension (degrees)
Sensory assessment of the upper limb | Single point of assessment at assessment day 1
  UL sensory testing using the Erasmus MC Modificatie van de (revised) Nottigham Sensory Assessment
Shoulder subluxation (palpation) | Single point of assessment at assessment day 1
  Palpating the gap between the acromion and the humeral head
Trunk control | Single point of assessment at assessment day 1
  Assessing the trunk impairment using the trunk impairment scale
Upper limb pain during walking | Single point of assessment at assessment day 1
  Using a numeric rating scale (0-10) to assess pain at the upper limb during walking
Gait speed | Single point of assessment at assessment day 1
  Calculating gait speed (m/s) based on the time it takes to complete the 10m walking

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium